CLINICAL TRIAL: NCT01351792
Title: A 12-week, Multicentre, Randomised, Double-blind, Double-dummy, 2-arm Parallel Group Study Comparing the Efficacy and Safety of Foster® 100/6 (Beclomethasone Dipropionate 100 µg Plus Formoterol 6 µg/Actuation), 2 Puffs b.i.d., Versus Symbicort® 200/6 (Budesonide 200 µg Plus Formoterol 6 µg/Actuation), 2 Inhalations b.i.d., on Parameters of Small Airway Function in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: A Study in Patients With Chronic Obstructive Pulmonary Disease (FAIR)
Acronym: FAIR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1007-PR-0045; 2010-022895-30 (EudraCT Number)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foster® (Experimental): Foster® (beclomethasone dipropionate 100 µg plus formoterol 6 µg/unit dose), 2 inhalations b.i.d. (daily dose of BDP "extrafine" 400 µg plus FF 24 µg).
  Interventions: Drug: Foster® 100/6 µg/unit dose
- Symbicort® Turbohaler® (Active Comparator): Symbicort® Turbohaler® (budesonide 200 μg plus formoterol fumarate 6 μg/actuation), 2 inhalations b.i.d. (daily dose of BUD 800 μg plus FF 24 μg).
  Interventions: Drug: Symbicort® Turbohaler® 200/6 μg/actuation

INTERVENTIONS:
Drug: Foster® 100/6 µg/unit dose — Foster® (beclomethasone dipropionate 100 µg plus formoterol 6 µg/unit dose), 2 inhalations b.i.d. (daily dose of BDP "extrafine" 400 µg plus FF 24 µg).
  Arms: Foster®
Drug: Symbicort® Turbohaler® 200/6 μg/actuation — Symbicort® Turbohaler® (budesonide 200 μg plus formoterol fumarate 6 μg/actuation), 2 inhalations b.i.d. (daily dose of BUD 800 μg plus FF 24 μg).
  Arms: Symbicort® Turbohaler®

SUMMARY:
The purpose of the present study is to demonstrate the higher efficacy of small particles Foster® 100/6 (two puffs b.i.d.) versus large particles Symbicort® 200/6 (two inhalations b.i.d.), in terms of residual volume reduction over a 12-week treatment period in Chronic Obstructive Pulmonary Disease (COPD) patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is an incurable, debilitating and progressive disease that can be fatal. The recent Global Burden of Disease Study ranks COPD as the 6th leading cause of mortality and the 12th leading cause of morbidity world-wide. Furthermore, trends in the use of medical care resources indicate that the economic cost of COPD continues to rise in direct relation to the ageing population, the increase in prevalence of disease and the cost of new and existing medical and public health interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 40 years, who have signed an Informed Consent form prior to initiation of any study-related procedure or when applicable written informed consent obtained by legal representative.
2. Outpatients with a clinical diagnosis of moderate to severe COPD and including:

   1. Smoking history of at least 10 pack years defined as [(number of cigarettes smoked per day) x (number of years of smoking)] / 20, both current and ex-smokers are eligible.
   2. Regular use of bronchodilators (e.g. β2-agonist, anticholinergics) in the 2 months before visit 1.
   3. Post-bronchodilator FEV1 < 65% of the predicted normal value at visit 1.
   4. Post-bronchodilator FEV1/FVC < 0.7 at visit 1.
   5. An increase in FEV1 < 15% and < 200 mL from baseline following administration of 400 µg of salbutamol at visit 1.
   6. Plethysmographic Functional Residual Capacity (FRC) > 120% of the predicted normal value (at visit 1 and visit 2).
   7. A Baseline Dyspnoea Index (BDI) focal score less or equal to 10 (at visit 1 and at visit 2).
3. A cooperative attitude and ability to be trained to the proper use of pMDI and DPI (Turbohaler®, inspiratory flow-driven, multidose powder inhaler) inhalers.

Main Exclusion Criteria:

1. Diagnosis of asthma or other clinically or functionally relevant respiratory disorders (other than COPD) which may interfere with data interpretation according to the investigator's opinion.
2. Clinically unstable concurrent disease: e.g. hyperthyroidism, diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; cardiovascular disease (e.g. coronary artery disease, hypertension, heart failure); gastrointestinal disease (e.g. active peptic ulcer); neurological disease; haematological disease; autoimmune disorders, or other which may impact the evaluation of the results of the study according to investigator's judgement.
3. Patients with COPD exacerbation and/or symptomatic infection of the airways requiring antibiotic therapy (at least 5 days) in the 2 months prior to screening and during the study period.
4. Patients treated with depot corticosteroids in the 2 months preceding the visit 1 and during the run-in period.
5. Major surgery in the previous 3 months and during the trial which may affect patient's compliance in study procedures (e.g. plethysmography).
6. Patients requiring chronic mechanical ventilation for COPD.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment in post-dose residual volume. | At day 84

SECONDARY OUTCOMES:
Changes from baseline in FEV1, FVC, FEV1/FVC, IVC/FVC, RV, TLC, RV/TLC, FRC, FRC/TLC, RV/VC, Raw, eff and sGaw, eff. | At day 84
Changes from baseline in airways resistance (R5, R20, R5-20) and reactance at 5 Hertz (X5) (in a subset of at least 50% of patients from pre-selected sites); | at day 84
Changes from baseline in COPD symptom scores (for each single score and the total score); | At day 84
Change from baseline in percentage of COPD symptom-free days; | At day 84
Change from baseline in rescue salbutamol or ipratropium bromide consumption (puffs per day); | At day 84
Change from baseline in percentage of rescue salbutamol or ipratropium bromide-free days; | At day 84
Transition Dyspnoea Index (TDI) score; | At day 84 (V4)
Clinical COPD Questionnaire (CCQ); | At screening (day -28), at baseline (day 0) and at the end of trial (day 84)
Physical activity (by means of pedometer); | Each day of the two weeks before each clinic visit
Nasal brushing (mRNA expression); | At screening (day -28), at baseline (day 0) and at the end of trial (day 84)
Number of patients with COPD exacerbations. | From pre-screening (day -35) to the end of trial (day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Dirkje Postma, MD, Study Chair — Dept. of Pulmonary Medicine and Tuberculosis - University of Groningen - The Netherlands; Marteen van den Berge, MD, Principal Investigator — Dept. of Pulmonary Medicine and Tuberculosis - University of Groningen - The Netherlands
Locations (1):
- Department of Pulmonary Diseases - University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Faiz A, Imkamp K, van der Wiel E, Boudewijn IM, Koppelman GH, Brandsma CA, Kerstjens HAM, Timens W, Vroegop S, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Steiling K, Spira A, Lenburg ME, Heijink IH, Postma DS, van den Berge M. Identifying a nasal gene expression signature associated with hyperinflation and treatment response in severe COPD. Sci Rep. 2020 Oct 15;10(1):17415. doi: 10.1038/s41598-020-72551-0. PMID 33060632
- [Derived] Boudewijn IM, Faiz A, Steiling K, van der Wiel E, Telenga ED, Hoonhorst SJM, Ten Hacken NHT, Brandsma CA, Kerstjens HAM, Timens W, Heijink IH, Jonker MR, de Bruin HG, Sebastiaan Vroegop J, Pasma HR, Boersma WG, Wielders P, van den Elshout F, Mansour K, Spira A, Lenburg ME, Guryev V, Postma DS, van den Berge M. Nasal gene expression differentiates COPD from controls and overlaps bronchial gene expression. Respir Res. 2017 Dec 21;18(1):213. doi: 10.1186/s12931-017-0696-5. PMID 29268739
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-022895-30